CLINICAL TRIAL: NCT01565213
Title: Transdiagnostic Group Treatments for Patients With Common Mental Disorders in Primary Health Care: A Randomized Controlled Trial
Brief Title: Transdiagnostic Group Treatments for Patients With Common Mental Disorders in Primary Health Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Kersti Ejeby, MD Head GP, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LS 0506-1010
Record Dates: First submitted 2012-03-19; First posted 2012-03-28 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Anxiety Disorders; Depressive Disorders; Stress Disorders
Keywords: primary health care,common mental disorders,; group therapy
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Stress Disorders, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CBT cognitive behavioral therapy (Active Comparator): group cognitive behavioural based therapy (CBT) administered by psychologists once a week for 12 weeks
  Interventions: Behavioral: CBT
- MMI Multimodal group intervention (Active Comparator): group multimodal intervention
  Interventions: Behavioral: MMI
- CAU (Other): Care as usual given by the GPs
  Interventions: Behavioral: CAU

INTERVENTIONS:
Behavioral: CBT — group cognitive behavioural based therapy (CBT) administered by psychologists once a week for 12 weeks,
  Arms: CBT cognitive behavioral therapy
Behavioral: MMI — group multimodal intervention (MMI) based on a protocol comprising a mix of existing group interventions and exercises borrowed from multiple techniques and therapeutic schools and administered by assistant nurses with brief training, including two sessions per week for 6 weeks.
  Arms: MMI Multimodal group intervention
Behavioral: CAU — Care as usual by the GPs
  Arms: CAU

SUMMARY:
The purpose of this study is to compare the effects of CBT and MMI on the quality of life and relief of psychological symptoms of patients with common mental disorders or problems attending primary health care centre.

DETAILED DESCRIPTION:
Design:

Clinical randomised non blinded controlled trial.

Setting:

The study was performed in an outpatient primary health care centre serving 36 000 inhabitants.

Participants:

Patients (n=278), aged 18-65 years, with common mental problems or disorders were referred to the study by the GPs and 245 were included in the study.

Interventions:

Participants were randomised to CAU or one of two group interventions in addition to CAU. These were: a) group cognitive behavioural based therapy (CBT) administered by psychologists once a week for 12 weeks, and b) group multimodal intervention (MMI) based on a protocol comprising a mix of existing group interventions and exercises borrowed from multiple techniques and therapeutic schools and administered by assistant nurses with brief training, including two sessions per week for 6 weeks.

Main outcome measures:

Primary outcome measure was the Mental Component Summary score of SF-36. Secondary outcome measures were perceived stress scale (PSS) and Self-Rating Scale for Affective Syndromes (CPRS-S-A)

ELIGIBILITY:
Inclusion Criteria:

* patients with common mental disorders or problems

Exclusion Criteria:

patients were excluded if:

* they met diagnostic criteria for bipolar or psychotic disorder or severe personality disorder,
* were judged to be at risk of committing suicidal acts, and
* if they had undergone MMI earlier. The investigators paid no consideration to whether patients were treated with SSRI medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2006-01; Primary Completion 2008-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change in Quality of life as measured by the SF-36 (Mental Component Score) | Change from baseline in SF-36 at 52 weeks

SECONDARY OUTCOMES:
Change in Psychopathology as measured by the Comprehensive Psychopathological Rating Scale Self-asssessmen (CPRS-S-A) | Change from baseline in CPRS-S-A at weeks 52

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Family and Community Medicine, Karolinska Institutet,, Huddinge, Sweden